CLINICAL TRIAL: NCT02230501
Title: Metabolic Activation With Protein-rich Formula Diet - a Randomized-controlled Trial
Brief Title: Metabolic Activation With Protein-rich Formula Diet
Acronym: AVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Almased Wellness GmbH (Industry)
Responsible Party: Principal Investigator, Stephan Martin, Principal investigator, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AVS
Record Dates: First submitted 2014-08-26; First posted 2014-09-03 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: For the second part of the study, i.e. the open-label registry, there ist no randomization.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: For the second part of the study, i.e. the open-label registry, 4000 subjects are anicipated.
Oversight: Data Monitoring Committee: No

ARMS (2):
- moderate diet regimen (Experimental): Week 1-4: replacement of breakfast and dinner with 1g PRMR /kg normal weight (=height in cm-100), a protein-rich lunch was allowed Week 5-12: replacement of dinner
  For this arm a local subgroup (n=55) and a nation-wide subgroup (n=100) is planned.
  Interventions: Dietary Supplement: moderate diet regimen
- stringent diet regimen (Experimental): Week 1: replacement of 3 main meals by 1g PRMR / kg normal weight (=height in cm - 100) Week 2-4: replacement of breakfast and dinner, a protein-rich lunch was allowed Week 5-12: replacement of dinner
  For this arm a local subgroup (n=55) and a nation-wide subgroup (n=100) is planned.
  Interventions: Dietary Supplement: stringent diet regimen

INTERVENTIONS:
Dietary Supplement: stringent diet regimen
  Other Names: protein-rich meal replacement (PRMR), i.e Almased-Vitalkost (Almased Wellness GmbH, Bienenbüttel, Germany)
  Arms: stringent diet regimen
Dietary Supplement: moderate diet regimen
  Other Names: protein-rich meal replacement (PRMR), i.e Almased-Vitalkost (Almased Wellness GmbH, Bienenbüttel, Germany)
  Arms: moderate diet regimen

SUMMARY:
Formerly, the investigators demonstrated in an uncontrolled proof-of principle study (NCT 01680926) that protein-rich meal replacement (PRMR) was successful in reducing daily insulin demand, HbA1c and weight in type 2 diabetes mellitus (T2DM) patients injecting >100 IE insulin/day. The aim of the present study was to investigate in a randomized-controlled trial if PRMR is also effective in T2DM patients treated with oral antidiabetic medication or insulin.

A second part of the study is an open-label registry for persons with type 2 diabetes, who will perform the lifestyle intervention with the stringent diet regime.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) patients had been randomized into two groups. During the 1st week the intervention group with stringent diet regime replaced 3 main meals by 50 g PRMR (Almased-Vitalkost, Almased Wellness GmbH, Bienenbüttel, Germany) each (=1100 kcal/day). In 2nd-4th week 2 meals were replaced and a protein-rich lunch was allowed. In 5th-12th week only dinner was replaced. The control group with moderate diet regime replaced breakfast and dinner for 4 weeks and then only dinner during the next 8 weeks. Clinical parameters were determined at the study center at baseline, after 4, 8 and 12 weeks. Primary endpoint was reduction of HbA1c, secondary endpoints reduction of weight and antidiabetic medication.

In the second part of the study type 2 diabetes patients are included in an open-label reistry and perform the lifestyle intervention with the stringent diet regime.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* HbA1c > 7,5%
* Body Mass Index (BMI) ≥ 27,5 kg/m2

Exclusion Criteria:

* acute infections
* severe diseased with hospital stay during the last 3 months
* chronic diseases
* chemotherapy or cortisone treatment
* weight loss of more than 2 kg per week during the last month
* smoking cessation during the last 3 months or planned
* weight-influencing medication
* pregnancy, breast-feeding or lack of contraception
* high-level physical activity of more than 1h per day
* incompatibility with components of the PRMR
* participation in an other study during the last 6 months

For the open-label registry, the only inclusion criterium is type 2 diabetes.

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  change in hemoglobin A1c

SECONDARY OUTCOMES:
HbA1c | 1 year
  change in hemoglobin A1c
body weight | 12 weeks and 1 year
  change in body weight
blood pressure | 12 weeks and 1 year
  change in systolic and diastolic blood pressure
cholesterol | 12 weeks and 1 year
  change in total cholesterol change in HDL cholesterol change in LDL cholesterol
fasting blood glucose | 12 weeks and 1 year
  change in fastin g blood glucose
quality of life | 12 weeks and 1 year
  change in SF-36 quality of life questionnaire change in ADS-L (German version of the general depression scale)
nutrition | 12 weeks and 1 year
  change in FEV (questionnaire for eating manners)
physical activity | 12 weeks and 1 year
  change in physical activity questionnaire
antidiabetic medication | 12 weeks and 1 year
  * absolute amount of antidiabetic medication
  * increase or reduction

CONTACTS AND LOCATIONS:
Locations (1):
- West German Centre of Diabetes and Health, Düsseldorf, Germany